# **Official Study Title:**

Optimizing Dimensions of Reinforcement to Enhance Behavioral Interventions

# **NCT Number:**

(To be assigned upon ClinicalTrials.gov registration)

**Document Type:** Informed Consent Form

# **Version Date:**

September 17, 2024

#### **Parental Permission to Participate in Research**

Translational Evaluation of Relapse Inoculation Procedures

#### Introduction

You are being asked to give permission for your child to participate in a research study that is being done by Dr. John Falligant, PhD who is an Assistant Professor in the Department of Psychological Sciences at Auburn University. This research is being conducted in collaboration with Dr. Michael Kranak at Oakland University.

Your decision to give permission for your child to participate in this study is voluntary. Your child does not have to be in this study. Your decision will not affect your or your child's present or future relationship with Auburn University, the researcher, or the Department of Psychological Sciences.

If you are an employee at Auburn University, your decision about your employment status. If you do not allow your child to participate in this project, there is no penalty or loss of benefits to you or your child at Auburn University.

# What is the purpose of this study?

The purpose of this research study is to analyze how individuals allocate their behavior between various response options given different types of rewards, magnitudes of rewards, and schedules of reinforcement.

# Who can participate in this study?

Your child is being asked to participate in the study because your child receives clinical services at Auburn University and they have demonstrated the pre-requisite skills required for this study (e.g., ability to follow simple instructions, attending skills).

#### How long will my child be in the study?

Sessions will be short (e.g., 5-10 minutes). Schedule permitting, we will run more than one session at a time. Your child's overall participation in this study should last no longer than 2-4 weeks.

#### Where will this study take place?

This study will take place within the Auburn University Center for Autism Research, Treatment, and Training (CARTT).

#### What will my child be asked to do?

Your child will be asked to your child will be asked to play games in which they will earn various preferred items (e.g., toys, snacks) based on how they respond to easy game tasks. The game will include simple tasks like matching, sorting, or pressing buttons and panels. The games will not interfere with your child's clinical treatment.

Game sessions may be recorded for data collection purposes. Only members of the research team will have access to the videos. They will be stored on a HIPAA- and FERPA-compliant cloud system (i.e., OneDrive).

Pseudonyms will be used for your child, this pseudonym will be your child's initials, which are already used within CARTT for HIPAA purposes.

# Are there any risks to my child?

There are no known research-related risks or discomforts.

With many research studies, there is a risk that someone who is not part of this research may accidentally see your child's personal information. Safeguards will be in place to minimize this risk by keeping your research records as confidential as possible. When the results of this research are published or presented at conferences, no information will be included that personally identifies your child.

### Are there any benefits to my child?

Although there may be no direct benefits to your child, the results of this study may benefit others in the future.

# Will I/my child receive anything for participating?

You/your child will not receive anything for participating in this study.

If your child is receiving medical treatment regardless of the research, no arrangements have been made for reimbursement for these procedures and you will be responsible for any expenses related to the treatment procedures. Please know that this research will **not** impact provision of clinical services.

# Who is the financial sponsor for this study?

The financial sponsor for this study is the National Institute of Child Health and Human Development (NICHD).

# Who could see my child's information?

Your child's research records may be shared and reviewed by the following groups:

- Representatives of the Oakland University Institutional Review Board (a collaborating site) and/or other regulatory compliance staff, whose job is to protect people who are in research studies.
- Regulatory authorities who oversee research (Office for Human Research Protections, or other federal, state, or international regulatory agencies)
- The financial sponsor supporting the study and their agents or monitors

De-identified data may be used or distributed to another investigator for future research use without additional permission from you.

# What if I/my child want to stop participating in this study?

If you/your child want to stop participating in this study, you/your child should contact the researcher because there may be special procedures to follow.

The researcher may stop your child's participation in this study at any time without your permission (e.g., pre-requisite skills not found to be present, or the study sessions no longer fit into the client's schedule). Should the research decide to terminate your child's participation, you will be contacted via email from the principal investigator.

# Who do I contact if I have questions about this study?

John Falligant, PhD Jmf0031@auburn.edu

For questions regarding your child's rights as a participant in human subject research, you may contact the Oakland University Institutional Review Board, 248-370-4898.

#### Signing the parental or legal guardian permission form

Your signature below means that you have read this form, or someone has read it to you, and you agree to give your child a permission to participate in the study.

| You are not giving up any legal rights by signing this pof this form. | parental permission form. You will be given a copy |
|---|---|
| Print name of participant/child | |
| Print name of parent or other person authorized to provide permission for participant/child | Signature of parent or other person authorized to provide permission for participant/child |
| Relationship to participant/child | Date |